CLINICAL TRIAL: NCT02995460
Title: Interval Training Study in Psoriatic Arthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: Helse Midt-Norge (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2012/1646
Record Dates: First submitted 2016-12-14; First posted 2016-12-16 (Estimated); Last update posted 2018-11-13 (Actual); Status verified 2018-11

CONDITIONS: Psoriatic Arthritis
Keywords: Exercise Therapy
MeSH Terms: conditions — Arthritis, Psoriatic | interventions — High-Intensity Interval Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- interval training (Experimental): 4x4 high intensity interval training was performed on a stationary bicycle with a supervisor twice a week and by one self-training a week.
  Interventions: Behavioral: interval training
- controls (No Intervention): No change in diet and training habits

INTERVENTIONS:
Behavioral: interval training — 4x4 high intensity interval training
  Arms: interval training

SUMMARY:
Psoriatic arthritis is a chronical inflammatory disease characterized by pain and reduced physical function. Patients have a higher risk of cardiovascular disease and a higher body mass index.

A pilot study in patients with rheumatoid arthritis has shown positive effect on inflammation after 12 weeks of high-intensity interval training.

The primary aim of this study is to determine whether high-intensity interval training affects the disease activity in psoriatic arthritis. This intervention is believed to result in benefits in terms of inflammation, body composition and risk factors for cardiovascular disease.

ELIGIBILITY:
Inclusion Criteria:

* fulfilling the CASPAR criteria of psoriatic arthritis
* ability to exercise.

Exclusion Criteria:

* Inability to exercise
* very high disease Activity
* unstable ischemic cardiovascular disease
* severe pulmonary disease
* pregnancy
* breastfeeding
* drug- and alcohol addictions

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Patient global assesment (PGA) | Baseline, 3 months (right after intervention), 9 months
  PGA is measured as a change between timepoints. PGA is registered by the patient on a visual analog scale.
Maximal oxygen uptake (VO2 max) | Baseline, 3 months (right after intervention), 9 months
  The VO2 max is measured as a change between timepoints

SECONDARY OUTCOMES:
Total lean mass | Baseline, 3 months (right after intervention), 9 months
  Total lean mass is measured as a change between timepoints and is measured by dual energy x-ray absorptiometry (DXA).
Total body fat | Baseline, 3 months (right after intervention), 9 months
  Total body fat is measured as a change between timepoints and is measured by dual energy x-ray absorptiometry (DXA).

CONTACTS AND LOCATIONS:
Overall Officials: Siri Forsmo, md prof, Study Director — Norwegian University of Science and Technology

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Thomsen RS, Nilsen TIL, Haugeberg G, Bye A, Kavanaugh A, Hoff M. Impact of High-Intensity Interval Training on Disease Activity and Disease in Patients With Psoriatic Arthritis: A Randomized Controlled Trial. Arthritis Care Res (Hoboken). 2019 Apr;71(4):530-537. doi: 10.1002/acr.23614. PMID 29882634
- [Result] Thomsen RS, Nilsen TIL, Haugeberg G, Bye A, Kavanaugh A, Hoff M. Effect of high-intensity interval training on cardiovascular disease risk factors and body composition in psoriatic arthritis: a randomised controlled trial. RMD Open. 2018 Oct 11;4(2):e000729. doi: 10.1136/rmdopen-2018-000729. eCollection 2018. PMID 30402265
- [Derived] Thomsen RS, Nilsen TIL, Haugeberg G, Sitter B, Kavanaugh A, Pedersen SJ, Hoff M. Changes of inflammation in patients with psoriatic arthritis after high intensity interval training assessed by ultrasound and MRI, a randomized controlled trial. BMC Musculoskelet Disord. 2023 Sep 19;24(1):743. doi: 10.1186/s12891-023-06871-3. PMID 37726677
- [Derived] Chronaiou I, Thomsen RS, Huuse EM, Euceda LR, Pedersen SJ, Hoff M, Sitter B. Quantifying bone marrow inflammatory edema in the spine and sacroiliac joints with thresholding. BMC Musculoskelet Disord. 2017 Nov 28;18(1):497. doi: 10.1186/s12891-017-1861-1. PMID 29179748